CLINICAL TRIAL: NCT06997523
Title: Effect of Breathing Therapy and Benson Relaxation Technique on Caregiver Burden, Perceived Stress and Self-Efficacy Among Alzheimer's Caregivers
Brief Title: Effects of Breathing Therapy and Benson Relaxation Technique on Caregivers of Alzheimer's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hülya Nuray Bayraktar (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Hülya Nuray Bayraktar, Graduate Student, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/12-01; 2024/23- 11
Record Dates: First submitted 2025-05-02; First posted 2025-05-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Caregiver Burden; Caregiver Stress; Caregiver; Caregiver Burden of People With Dementia; Self Efficacy
Keywords: Alzheimer; Caregiver; Self Efficacy; Stress; Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Intervention Group will be given breathing therapy and Benson relaxation technique training for 6 weeks.
  Interventions: Behavioral: Breath Therapy and Benson Relaxation Technique
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Breath Therapy and Benson Relaxation Technique — Relaxing breathing therapy (4-7-8) and Benson relaxation technique will be applied to the intervention group for 6 weeks. No intervention will be made to the control group.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of respiratory therapy and the Benson Relaxation Technique on caregiver burden, perceived stress, and self-efficacy among caregivers of individuals with Alzheimer's disease. The study will be conducted at the Geriatrics Outpatient Clinic of Gülhane Training and Research Hospital, University of Health Sciences, between February and May 2025. A total of 80 healthy adult caregivers aged 18 to 65 will be enrolled and randomly assigned to either the intervention group (n=40) or the control group (n=40). The intervention group will participate in a structured 6-week program consisting of face-to-face group sessions with a maximum of 10 participants per group, held twice weekly. Each 30-minute session will include 10 minutes of guided respiratory therapy followed by 20 minutes of the Benson Relaxation Technique. The control group will receive routine care without any additional interventions. The purpose of this study is to evaluate whether the combined application of respiratory therapy and the Benson Relaxation Technique results in significant improvements in caregiver outcomes. Caregivers will be assessed using standardized measures, including the Caregiver Burden Scale for Dementia, the Perceived Stress Scale, and the General Self-Efficacy Scale. Assessments will be conducted at baseline (week 0), week 2, week 4, week 6 (end of intervention), and week 8 (two weeks post-intervention). The study is guided by the following hypotheses: H01: Respiratory therapy and the Benson Relaxation Technique have no effect on caregiver burden. H11: Respiratory therapy and the Benson Relaxation Technique reduce caregiver burden. H02: Respiratory therapy and the Benson Relaxation Technique have no effect on perceived stress. H12: Respiratory therapy and the Benson Relaxation Technique reduce perceived stress. H03: Respiratory therapy and the Benson Relaxation Technique have no effect on self-efficacy. H13: Respiratory therapy and the Benson Relaxation Technique improve self-efficacy.

DETAILED DESCRIPTION:
The intervention in this study consists of two evidence-based non-pharmacological techniques: the 4-7-8 relaxing breathing technique and the Benson Relaxation Technique. These methods were delivered in a structured format over six weeks to support caregivers of individuals diagnosed with Alzheimer's disease. The 4-7-8 breathing technique is a rhythmic breathing practice designed to induce physiological calm by modulating the autonomic nervous system. The specific procedure followed was:

* Participants were seated comfortably with a straight posture and used provided eye masks to minimize visual distractions.
* The tongue was placed behind the upper front teeth and maintained in this position throughout the exercise.
* A full exhalation was performed through the mouth while producing a soft whooshing sound.
* This was followed by a quiet nasal inhalation for 4 seconds, breath-holding for 7 seconds, and a controlled exhalation through the mouth over 8 seconds.
* This cycle was repeated approximately three times per minute, totaling 30 cycles in a 10-minute session.

The Benson Relaxation Technique, widely used in mind-body therapy, aims to elicit the relaxation response through passive focus and muscular relaxation. The steps included:

* Selecting a personal word or phrase (e.g., "peace," "health," "love") to silently repeat during exhalation.
* Sitting quietly with eyes closed, participants gradually relaxed all major muscle groups from feet to head.
* While breathing naturally, they repeated the chosen word silently on each exhalation.
* A passive attitude was encouraged; distracting thoughts were acknowledged and released without judgment, redirecting attention to the breath and word.
* Sessions concluded with a quiet reorientation period before standing. Inclusion criteria: Adults aged 18-65 who were the primary caregivers of individuals diagnosed with Alzheimer's disease for at least six months; at least primary school graduates; cognitively and physically able to perform the exercises and complete forms; and provided informed consent.

Exclusion criteria: Individuals with psychological disorders (e.g., anxiety, depression), advanced cardiac, pulmonary (e.g., COPD, asthma), or oncological conditions; communication impairments (vision, hearing, or speech); those undergoing hospitalization or surgery during the study period; or those already engaged in other structured relaxation methods such as yoga or meditation.

Rationale: Caregivers of Alzheimer's patients frequently experience chronic stress and burden, leading to emotional exhaustion, physical health issues, and reduced quality of life. Breathing-based and meditative interventions offer accessible, cost-effective strategies to counteract these effects and improve psychological resilience.

Study Design Notes:

* This is a randomized, controlled.
* Participants were assigned to groups using a computer-based randomization tool.
* All sessions were held face-to-face in groups of ≤10 participants, and all interventions were delivered by the same researcher to ensure standardization.

This structured intervention model was designed to provide both physiological relaxation (via controlled breathing) and psychological relief (via cognitive disengagement and passive awareness), aiming to support caregiver well-being through an integrative mind-body approach.

Statistical Analysis: Data were analyzed using SPSS version 23.0. Groups were anonymized as "A" and "B". Normality was evaluated via Shapiro-Wilk test, skewness-kurtosis values, and Q-Q plots. Parametric tests (Student's t-test, paired samples t-test, ANOVA) were used for normally distributed data, while non-parametric tests (Mann-Whitney U, Friedman) were applied otherwise. Categorical variables were analyzed using chi-square tests. Descriptive statistics included means ± SD or medians (min-max). Cronbach's alpha was calculated for scale reliability. A p-value <0.05 was considered statistically significant.

This study received ethical approval from the Hacettepe University Clinical Research Ethics Committee under approval numbers 2024/12-01 and 2024/23-11, dated June 26, 2024, and December 3, 2024, respectively. Additionally, regulatory approval was obtained from the Turkey Medicines and Medical Devices Agency with decision number E-85521274-000-3587573 dated January 16, 2025. All participants provided written informed consent prior to participation. Confidentiality and data security were strictly maintained throughout the study to protect participant privacy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* At least primary school graduate
* First degree caregiver of a patient diagnosed with Alzheimer's (continuous caregiver, family member, spouse, etc., or paid continuous caregiver)
* Caring for an individual diagnosed with Alzheimer's for at least 6 months
* Cognitively and physically capable of answering data collection forms and implementing the taught exercise with the researcher Caregivers who agree to participate in the study will be included in the sample.

Exclusion Criteria:

* Individuals with cognitive and psychological problems (anxiety, panic attacks, depression, etc.)
* Those diagnosed with advanced heart disease, asthma, COPD, and advanced cancer
* Those with communication problems (hearing, vision, speech, etc.)
* Individuals who are hospitalized or undergo surgery, etc. during the study period
* Individuals who are simultaneously continuing another relaxation exercise (yoga, meditation, visualization, etc.) will not be included in the sample.

In addition, caregivers who indicate that they want to withdraw from the study during the study and who do not attend the weekly group sessions twice in a row will be excluded from the sample.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden as measured by the Caregiver Burden Scale for Dementia | Assessed at baseline (week 0), week 2, week 4, week 6 (end of intervention)
  Caregiver burden will be assessed using the Caregiver Burden Scale for Dementia, which includes four sub-dimensions: physical, social, economic, and psychological. The scale consists of 24 items, each rated on a 5-point Likert scale ranging from 1 ("Never") to 5 ("Always"). There are no reverse-coded items. The total score ranges from 24 to 120, with higher scores indicating a greater caregiver burden. Subscale scores and total scores will be compared between the intervention and control groups at each assessment point to evaluate changes over time.
Change in Perceived Stress as Measured by the Perceived Stress Scale | Assessed at baseline (week 0), week 2, week 4, week 6 (end of intervention)
  Perceived stress will be assessed using the Perceived Stress Scale for Adults. This scale consists of 14 items designed to measure the degree to which situations in one's life are appraised as stressful. Items are rated on a 5-point Likert scale from 0 ("Never") to 4 ("Very Often"). Items 4, 5, 6, 7, 9, 10, and 13 are reverse-scored. Total scores range from 0 to 56, with higher scores indicating greater levels of perceived stress. Changes in perceived stress will be evaluated by comparing scores at different time points within and between groups.
Change in Self-Efficacy as Measured by the General Self-Efficacy Scale | Assessed at baseline (week 0), week 2, week 4, week 6 (end of intervention)
  Self-efficacy will be assessed using the General Self-Efficacy Scale, which includes 10 items aimed at measuring an individual's belief in their ability to cope with a variety of difficult demands. Each item is rated on a 4-point Likert scale ranging from 1 ("Not at all true") to 4 ("Exactly true"). Total scores range from 10 to 40, with higher scores reflecting greater perceived self-efficacy. Group differences and within-group changes over time will be analyzed.

SECONDARY OUTCOMES:
Change in Caregiver Burden Two Weeks After the Intervention as Measured by the Caregiver Burden Scale for Dementia | From week 6 to week 8
  Caregiver burden will be assessed using the Caregiver Burden Scale for Dementia, which includes four sub-dimensions: physical, social, economic, and psychological. The scale consists of 24 items, each rated on a 5-point Likert scale ranging from 1 ("Never") to 5 ("Always"). There are no reverse-coded items. The total score ranges from 24 to 120, with higher scores indicating a greater caregiver burden. Subscale scores and total scores will be compared between the intervention and control groups at each assessment point to evaluate changes over time.
Change in Perceived Stress Two Weeks After the Intervention as Measured by the Perceived Stress Scale | From week 6 to week 8
  Perceived stress will be assessed using the Perceived Stress Scale for Adults. This scale consists of 14 items designed to measure the degree to which situations in one's life are appraised as stressful. Items are rated on a 5-point Likert scale from 0 ("Never") to 4 ("Very Often"). Items 4, 5, 6, 7, 9, 10, and 13 are reverse-scored. Total scores range from 0 to 56, with higher scores indicating greater levels of perceived stress. Changes in perceived stress will be evaluated by comparing scores at different time points within and between groups.
Change in Self-Efficacy Two Weeks After the Intervention as Measured by the General Self-Efficacy Scale | From week 6 to week 8
  Self-efficacy will be assessed using the General Self-Efficacy Scale, which includes 10 items aimed at measuring an individual's belief in their ability to cope with a variety of difficult demands. Each item is rated on a 4-point Likert scale ranging from 1 ("Not at all true") to 4 ("Exactly true"). Total scores range from 10 to 40, with higher scores reflecting greater perceived self-efficacy. Group differences and within-group changes over time will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Nuray Bayraktar, Master's Stu, Principal Investigator
Locations (1):
- Gulhane Training and Education Hospital, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No